CLINICAL TRIAL: NCT05985109
Title: A Phase II Multi-cohort Clinical Study Evaluating The Efficacy and Safety of KN046 in Combination With Regorafenib for Metastatic Microsatellite-Stable Colorectal Cancer: a Phase II Multi-cohort Study
Brief Title: KN 046 Plus Regorafenib in MSS Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGOG-KREC-01
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-liver metastasis cohort (Experimental): Arm A will include microsatellite-stable metastatic colorectal cancer patients who have no active liver metastasis. Patients are required to have received prior 5-Fu， oxaliplatin, and irinotecan treatment before enrollment.
  Interventions: Drug: KN046; Drug: regorafenib
- BRAF V600E mutant cohort (Experimental): Arm B will include microsatellite-stable metastatic colorectal cancer patients who have BRAF V600E mutation. Patients are required to have received prior 5-Fu， oxaliplatin, and irinotecan treatment before enrollment.
  Interventions: Drug: KN046; Drug: regorafenib
- Front-line therapy cohort (Experimental): Arm C will include microsatellite-stable metastatic colorectal cancer patients who are unable or refuse to receive standard first-line or second-line treatment.
  Interventions: Drug: KN046; Drug: regorafenib

INTERVENTIONS:
Drug: KN046 — KN046 is a recombinant humanized PD-L1/CTLA-4 bispecific single-domain antibody that blocks both PD-L1 interaction with PD-1 and CTLA-4 interaction with CD80/CD86.
Drug: regorafenib — Regorafenib is a multi-target tyrosine kinase inhibitors and is one of the standard third-line therapy in mCRC

SUMMARY:
The study is an interventional Phase II clinical trial aiming to optimize immunotherapy strategies for microsatellite-stable colorectal cancer. We will include three types of metastatic colorectal cancer patients: those without liver metastasis, or carrying BRAF V600E mutation, or unable to tolerate chemotherapy as their initial or second-line treatment. The participants will receive a combination treatment of regorafenib and KN046 which is a PD-L1/CTLA-4 bispecific antibody. Treatment efficacy and safety profile would be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

I01. Subjects are able to comprehend the informed consent form, voluntarily participate, and sign the informed consent form.

I02. Subjects are ≥18 years old on the day of signing the informed consent form, with no gender restrictions.

I03. Histologically confirmed colorectal adenocarcinoma, including signet ring cell carcinoma and mucinous adenocarcinoma.

I04. According to RECIST 1.1 criteria, there should be at least one measurable or evaluable lesion at baseline. If the subject has only one measurable or evaluable lesion at baseline, the lesion must not have been exposed to radiotherapy previously, or there must be evidence of significant progression after radiotherapy treatment completion.

I05. ECOG performance status of 0 or 1. I06. Expected survival ≥3 months. I07. Archived tumor tissue samples or freshly obtained tumor tissue samples are available.

I08. Female subjects of childbearing potential or male subjects with partners of childbearing potential agree to use highly effective contraception from 7 days before the first dose until 120 days after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose.

I09. Subjects have the ability and willingness to comply with the study protocol's visits, treatment plan, laboratory tests, and other study-related procedures.

I10. Within the first 7 days of initial dosing, subjects should have good organ function:

HGB ≥ 80g/L NEU ≥ 1.0*10^9/L PLT ≥ 75*10^9/L Cr≤1.5×ULN or CrCl≥50mL/min（ Cockcroft-Gault method） TBiL ≤ 1.5×ULN ALT and AST ≤3 ×ULN； for patients with liver metastasis ALT and AST ≤5 ×ULN urine protein <2+；if urine protein ≥ 2+，24 hour urinary protein quantity <2g； INR， APTT，PT ≤ 1.5 ×ULN

I11. For each cohort, the previous treatment history must meet the following conditions:

Cohort A: pMMR/MSS mCRC with no BRAF V600E mutation, who failed fluoropyrimidine, oxaliplatin, and irinotecan treatments, and without definitive active liver metastases at enrollment (judged by the investigator based on medical history and imaging).

Cohort B: pMMR/MSS mCRC with BRAF V600E mutation, who failed fluoropyrimidine, oxaliplatin, and irinotecan treatments.

Cohort C: MSS mCRC that has not intolerant or unsuitable for or refuse to receive standard first-line or second-line chemotherapy.

Exclusion Criteria:

E01. Subjects with untreated active brain metastases or meningeal metastases; if the subject's brain metastases have been treated and the metastases are stable (brain imaging at least 4 weeks before the first dose shows stable lesions, and there is no evidence of new neurological symptoms or the neurological symptoms have returned to baseline), then enrollment is allowed.

E02. Subjects with a history of gastrointestinal perforation or fistula within 6 months before the first dose. If the perforation or fistula has been treated with resection or repair, and the disease is judged to be recovered or improved by the investigator, then enrollment is allowed.

E03. Subjects who have received any other interventional clinical trial or any other antitumor treatment within 28 days or 5 half-lives before the first dose (whichever is shorter). Palliative radiotherapy for bone metastases to relieve symptoms is permitted.

E04. Subjects who have undergone major surgery within 28 days before the first dose (e.g., major abdominal or thoracic surgery; excluding drainage, diagnostic puncture, or peripheral vascular access replacement).

E05. Subjects who require systemic corticosteroids (≥10 mg/day prednisone or equivalent) or immunosuppressive therapy for a continuous 7-day period within 14 days before the first dose. Inhaled or locally applied steroids and physiological replacement doses of steroids due to adrenal insufficiency are allowed. Short-term (≤7 days) corticosteroids for prophylaxis (e.g., contrast dye allergy) or treatment of non-autoimmune diseases (e.g., delayed hypersensitivity reaction caused by exposure to allergens) are allowed.

E06. Subjects who have received live vaccines (including attenuated live vaccines) within 28 days before the first dose.

E07. Subjects with interstitial lung disease or a history of non-infectious pneumonia requiring oral or intravenous corticosteroid treatment.

E08. Subjects with active autoimmune diseases requiring systemic treatment within 2 years before the start of the study or those considered at risk of recurrence or planned treatment for autoimmune diseases as judged by the investigator. Exclusions include a) skin diseases that do not require systemic treatment (e.g., vitiligo, alopecia, psoriasis, or eczema); b) hypothyroidism caused by autoimmune thyroiditis, requiring stable doses of hormone replacement therapy; c) type 1 diabetes requiring stable doses of insulin replacement therapy; d) childhood asthma fully resolved with no need for intervention in adulthood; e) the investigator judges that the disease will not relapse without external triggering factors.

E09. Subjects with a history of other malignant tumors within 5 years, excluding cured skin squamous cell carcinoma, basal cell carcinoma, non-invasive bladder carcinoma, localized low-risk prostate cancer (defined as stage ≤T2a, Gleason score ≤6, and prostate-specific antigen (PSA) ≤10 ng/mL (if measured) in patients who have undergone curative treatment and have no biochemical recurrence of prostate-specific antigen (PSA)), in situ cervical/breast carcinoma, or Lynch syndrome.

E10. Subjects with uncontrolled comorbidities, including but not limited to: a) active HBV or HCV infection; b) subjects who are HBsAg positive and/or HCV antibody positive during screening must undergo HBV DNA and/or HCV RNA testing. Only subjects with HBV DNA ≤500 IU/mL (or ≤2000 copies/mL) and/or HCV RNA negative can be enrolled; HBV DNA monitoring will be at the discretion of the investigator based on the subject's condition during the trial; c) known HIV infection or AIDS history; d) active tuberculosis; e) active infection or systemic use of anti-infective drugs for more than 1 week within 28 days before the first dose; fever of unknown cause within 2 weeks before the first dose; f) uncontrolled hypertension (resting blood pressure ≥160/100 mmHg), symptomatic congestive heart failure (NYHA II-IV), unstable angina or myocardial infarction within 6 months, or the presence of QTc prolongation or the risk of arrhythmia (baseline QTc >470 msec <Fridericia method correction>, difficult-to-correct hypokalemia, long QT syndrome, atrial fibrillation with resting heart rate >100 bpm, or severe valvular heart disease); g) active bleeding that cannot be controlled after medical treatment.

E11. Toxicity from previous antitumor treatments has not recovered to Grade ≤2 (NCI-CTCAE v5.0) or baseline, except for alopecia, skin pigmentation (allowed at any level), and immune-related adverse reactions requiring physiological replacement (e.g., hypothyroidism, hypopituitarism, type 1 diabetes).

E12. History of allogeneic bone marrow or organ transplantation. E13. Previous history of allergic reactions, hypersensitivity reactions, or intolerance to antibody drugs (e.g., severe allergic reactions, immune-mediated hepatotoxicity, immune-mediated thrombocytopenia, or anemia).

E14. Pregnant and/or lactating females. E15. Other conditions that, in the investigator's opinion, may affect the safety or compliance of the study drug treatment, including but not limited to moderate to large pleural/ascites/pericardial effusion, uncorrectable pleural/ascites/pericardial effusion, intestinal obstruction or subacute intestinal obstruction, psychiatric disorders, etc.

E16. Previous treatment with any immune checkpoint inhibitors or T-cell co-stimulatory drugs, including but not limited to PD-1/PD-L1, CTLA-4, LAG3, and other immune checkpoint inhibitors, therapeutic vaccines, etc.

E17. Previous treatment with regorafenib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Objective response rate (defined as CR+PR) will be reported based on investigator's evaluation.

SECONDARY OUTCOMES:
Disease control rate | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Disease control rate (defined as CR+PR+SD) will be reported based on investigator's evaluation.
Progression free survival | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Progression-free survival (PFS) is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic progressive disease (PD) or death due to any cause.
Duration of response | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Duration of response (DOR) is defined as the time from the date of the first response to the first objective documentation of radiographic progressive disease (PD) or death due to any cause.
Overall survival | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Overall survival (OS) is defined as the time from the date of first dose to the date of death from any cause.
treatment-related adverse event | Informed consent to 30 days after last dose of treatment
  A treatment-related adverse event (TRAE) is defined as any adverse event not present prior to the initiation of drug treatment or any adverse event already present that worsens in intensity or frequency following exposure to the drug treatment. TRAEs were graded using National Cancer Institute (NCI)-CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No